CLINICAL TRIAL: NCT02415257
Title: Gentamicin Treatment Prior to Vestibular Schwannoma Surgery in Patients With no Measurable Remaining Vestibular Function
Brief Title: Gentamicin Treatment Prior to Schwannoma Surgery - No Residual Function
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VS-FT-02
Record Dates: First submitted 2015-01-26; First posted 2015-04-14 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Vestibular Schwannoma
Keywords: Vestibular schwannoma; acoustic neuroma; cerebellopontine angle tumour; gentamicin; rehabilitation; postural balance
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gentamicin treated (Experimental): Installation of gentamicin in the middle ear 6 weeks prior to surgery + rehabilitation exercises before and after both treatment and surgery.
  Rehabilitation exercises are not considered to be an intervention since their benign impact on vestibular/postural compensation is well documented and exclusion from exercises would not be approved by the ethical board
  Interventions: Drug: Gentamicin
- Non-gentamicin (No Intervention): Rehabilitation exercises before and after both treatment and surgery Rehabilitation exercises are not considered to be an intervention since their benign impact on vestibular/postural compensation is well documented and exclusion from exercises would not be approved by the ethical board

INTERVENTIONS:
Drug: Gentamicin — Intratympanic installation of gentamicin 2-4 times depending on the efficacy of vestibular deafferentation
  Other Names: prehabituation
  Arms: Gentamicin treated

SUMMARY:
The purpose of the study is to determine whether vestibular and postural compensation following schwannoma surgery is improved by ablating vestibular function prior to surgery, even if vestibular function is absent according to modern assessment techniques

DETAILED DESCRIPTION:
Patients subjected to vestibular schwannoma surgery most often suffer from vertigo after surgery, even if no vestibular function can be found in pre-surgical assessment. According to retrospective data about 33% of patients scheduled for surgery do not have any measurable vestibular function. Even the occurrence of spontaneous nystagmus has been recorded in patients with no or very little function prior to surgery (Parietti-Winkler et al. 2008 JNNP). This indicates that despite new methods of measuring vestibular function, remaining vestibular function can be present and patients might benefit from pre-treatment of gentamicin (Tjernström et al. 2009 JNNP)

ELIGIBILITY:
Inclusion Criteria:

* Vestibular schwannoma advised to surgical treatment
* No measurable remaining vestibular function

Exclusion Criteria:

* impaired decision making
* neurofibromatosis
* signs for central dysfunction
* remaining vestibular function
* Patients are advised not to participate in the gentamicin arm if
* hearing is better than 30 deciBel (dB) in pure tone average (500, 1000, 2000, 3-4000 Hz) and speech discrimination better than 70%
* the neurosurgeon aim at hearing preservation surgery and do not want to risk gentamicin associated hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Differences and changes of postural control following surgery, compared to before surgery | At first vestibular assessment at the time for inclusion and 6 months after surgery
  Postural control assessed with posturography during a sensory conflict

SECONDARY OUTCOMES:
Occurrence of spontaneous nystagmus after surgery | Day 1 after surgery and for the duration of either spontaneous nystagmus or hospital stay (up to 2 weeks)
  To measure spontaneous nystagmus and its direction after surgery as a sign of vestibular deafferentation or central nervous damage
Change of hearing levels | At first vestibular assessment and 4weeks after gentamicin installation
  Measuring hearing levels (pure tone average and speech discrimination) before and after gentamicin treatment to determine possible detrimental effects on hearing
Differences in the level of stress after surgery | Daily after surgery for the duration of the hospital stay, up to 2 weeks
  Measuring cortisol in the saliva after surgery during the time patients are admitted to the hospital
Differences of subjective well being after surgery | Immediate time after surgery (2weeks)
  Daily subjective assessment of perceived vertigo/dizziness after surgery
Differences of duration of hospital stay | After surgery for the duration of the hospital stay up to 2 weeks
  Length of hospital stay required before patients can be discharged
Differences of subjective well being after gentamicin treatment | Immediate time after gentamicin treatment (2weeks)
  Daily subjective assessment of perceived vertigo/dizziness after gentamicin treatment
Differences of perceived dizziness after surgery | 6 months after surgery
  Measurement of level of dizziness in daily life, questionnaire Dizziness Handicap Inventory (DHI)
Differences of perceived anxiety/depression after surgery | 6 months after surgery
  Measurement of level of anxiety/depression in daily life, questionnaire Hospital Anxiety and Depression Scale (HADS)
Change of level of perceived dizziness after surgery as compared to before surgery | At first vestibular assessment (inclusion) and 6 months after surgery
  Measurement of level of dizziness in daily life, questionnaire Dizziness Handicap Inventory (DHI)
Change of level of perceived anxiety/depression after surgery as compared to before surgery | At first vestibular assessment (inclusion) and 6 months after surgery
  Measurement of level of anxiety/depression in daily life, questionnaire Hospital Anxiety and Depression Scale (HADS)
Differences in vestibular compensation after surgery | 6 months after surgery
  Vestibular function tests; v-HIT (head impulse test), calorics and otolith tests to determine compensation and function after surgery
Change of vestibular function after gentamicin treatment | 6 weeks after gentamicin treatment
  Vestibular function tests; v-HIT (head impulse test), calorics and otolith tests to determine compensation and function after gentamicin treatment

OTHER OUTCOMES:
Differences of needed sick-leave from work and leisure activities | 6 months after surgery
  Time for return to normal daily activities after surgery, both job-related and leisure.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Tjernström, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Dept. OtoRhinoLaryngology Head and Neck Surgery, Skane University Hospital, Lund, Sweden

REFERENCES:
- [Background] Parietti-Winkler C, Gauchard GC, Simon C, Perrin PP. Visual sensorial preference delays balance control compensation after vestibular schwannoma surgery. J Neurol Neurosurg Psychiatry. 2008 Nov;79(11):1287-94. doi: 10.1136/jnnp.2007.135913. Epub 2008 Aug 1. PMID 18676407
- [Background] Magnusson M, Padoan S. Delayed onset of ototoxic effects of gentamicin in treatment of Meniere's disease. Rationale for extremely low dose therapy. Acta Otolaryngol. 1991;111(4):671-6. doi: 10.3109/00016489109138398. PMID 1950529
- [Result] Tjernstrom F, Fransson PA, Kahlon B, Karlberg M, Lindberg S, Siesjo P, Magnusson M. Vestibular PREHAB and gentamicin before schwannoma surgery may improve long-term postural function. J Neurol Neurosurg Psychiatry. 2009 Nov;80(11):1254-60. doi: 10.1136/jnnp.2008.170878. Epub 2009 Jul 1. PMID 19574236
- [Result] Magnusson M, Kahlon B, Karlberg M, Lindberg S, Siesjo P, Tjernstrom F. Vestibular "PREHAB". Ann N Y Acad Sci. 2009 May;1164:257-62. doi: 10.1111/j.1749-6632.2009.03778.x. PMID 19645909
- [Result] Magnusson M, Karlberg M, Tjernstrom F. 'PREHAB': Vestibular prehabilitation to ameliorate the effect of a sudden vestibular loss. NeuroRehabilitation. 2011;29(2):153-6. doi: 10.3233/NRE-2011-0689. PMID 22027076
- [Result] Magnusson M, Kahlon B, Karlberg M, Lindberg S, Siesjo P. Preoperative vestibular ablation with gentamicin and vestibular 'prehab' enhance postoperative recovery after surgery for pontine angle tumours--first report. Acta Otolaryngol. 2007 Dec;127(12):1236-40. doi: 10.1080/00016480701663433. PMID 17917842